CLINICAL TRIAL: NCT02519309
Title: Dietary Intervention in Type-2 Diabetics and Pre-Diabetics Emphasizing Personalized Carbohydrate Intake
Brief Title: Dietary Intervention in Type-2 Diabetes and Pre-Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virta Health (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1
Record Dates: First submitted 2015-08-04; First posted 2015-08-10 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 2; Pre-diabetes; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: 1. open label, non-randomized, before-and-after study of patients with type 2 diabetes who self-select the intervention (with education delivered via onsite group classes or web-based, self-selected by participant) or usual care
  2. single arm, before-and-after study of patients with prediabetes who self-select to receive the intervention (no comparison group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- onsite (Experimental): Education (the virta program) for the onsite group will be delivered in person, with 26 classes over 12 months including group and individual sessions. Sessions will be scheduled weekly for the first 3 months, biweekly during months 4-6, and monthly thereafter. Each session will last approximately 90 minutes.
  Interventions: Other: Virta Program
- web-based (Experimental): Education (the virta program) for the web-based educational group will be the same content as the onsite group, but delivered via the web and completed at the participant's own pace.
  Interventions: Other: Virta Program
- Control (usual care) (No Intervention): The study will make no intervention to this group. Participants in this group will be recent referrals to a local diabetes education program and care for their condition will continue to be managed by their own medical providers.

INTERVENTIONS:
Other: Virta Program
  Arms: onsite; web-based

SUMMARY:
The primary purpose of this research is to demonstrate the therapeutic effects of implementing a well-formulated low carbohydrate lifestyle program over 2 years in patients with type 2 diabetes, pre-diabetes, and metabolic syndrome.

DETAILED DESCRIPTION:
The primary purpose of this research is to demonstrate the therapeutic effects of implementing a well-formulated low carbohydrate lifestyle program over 2 years. Positive therapeutic effects would be represented by improved glycemic control in patients with type 2 diabetes without use of additional glycemic control medications and failure to progress to type 2 diabetes in individuals with pre-diabetes and metabolic syndrome.

Secondary purposes of this research are to determine if therapeutic effects of the intervention differ between patients who self-select onsite vs. web-based education delivery, explore relationships between change in LDL cholesterol and carotid intima media thickness, and to evaluate the sustainability of health outcomes achieved and the economic impact of therapeutic effects over 5 years.

ELIGIBILITY:
Inclusion Criteria:

Body weight/Diabetes:

* Diagnosis of type-2 diabetes with BMI > 25 (without end-organ failure)
* Fasting glucose >126 mg/dL or HbA1c >6.5

Body weight/ Pre-diabetes:

• Diagnosis of metabolic syndrome with BMI >30 and HbA1c > 5.6 (note: this does not apply to usual care control subjects)

Ethnicity: all ethnic groups

Exclusion Criteria:

* BMI <30 without diagnosis of Type-2 diabetes, metabolic syndrome
* Type 1 diabetes
* History of keto-acidosis
* History of MI, stroke, angina, coronary insufficiency within the last 6 months
* Diabetic retinopathy requiring treatment
* Creatinine > 2.0
* Urinary albumin > 1 g/d
* Impaired hepatic function (Bilirubin >2, Albumin < 3.5)
* Cholelithiasis or biliary dysfunction
* Cancer requiring treatment in the past 5 years, with the exception of non-melanoma skin cancer
* Chronic infectious disease requiring ongoing treatment
* Other chronic diseases or condition likely to limit lifespan to <6 years
* Non-English speaking
* Unable or unwilling to participate in group sessions (e.g., plans to relocate within the next year) or conform to a carbohydrate restricted diet lifestyle (e.g., food intolerances, religious or personal restrictions)
* Weight loss of >10% in past 6 months
* Currently pregnant or nursing, or planning to become pregnant during the study
* Major psychiatric disorder (e.g., schizophrenia, bipolar disorder) currently uncontrolled
* Excessive alcohol intake (acute or chronic) defined as average consumption of 3 or more alcohol-containing beverages daily or consumption of more than 14 alcoholic beverages per week

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Type-2 Diabetes Status | 3 Months (intervention arms only), 12 and 24 Months (intervention and usual care arms)
  Type-2 diabetes status will be evaluated by measuring Hemoglobin A1c (HbA1c)
Change from Baseline Metabolic Syndrome Status | 3 Months (intervention arms only), 12 and 24 Months (intervention and usual care arms)
  Metabolic syndrome status will be evaluated by standard markers. Metabolic syndrome is defined as having at least three of the following:
  * Waist circumference: ≥40 inches (men) or ≥35 inches (women)
  * Fasting triglycerides: ≥150 mg/dL
  * HDL-C: <40 mg/dL (men) or <50 mg/dL (women)
  * Blood pressure: ≥130/85 mm Hg or use of hypertensive medication
  * Fasting glucose: ≥ 100 mg/dL or use of hyperglycemia medication
Change from Baseline Body Weight | 3 Months (intervention arms only), 12 and 24 Months (intervention and usual care arms)
  Body weight will be evaluated on a calibrated scale

SECONDARY OUTCOMES:
Change from Baseline Carotid Intima Media Thickness (CIMT) (intervention and usual care arms, participants with type 2 diabetes only) | 12 and 24 Months
  Ultrasound Measurement of the Carotid Artery
Change from Baseline Serum Lipids | 3 Months (intervention arms only), 12 and 24 Months (intervention and usual care arms)
  Serum lipids including lipoprotein size and number
Change from Baseline Body Composition | 3,12 and 24 Months (intervention arms only)
  Body composition will be determined using dual-energy X-ray absorptiometry (DXA), which provides accurate information on total body and regional fat, lean body mass, and bone mass
Change from Baseline Type-2 Diabetes Status | 42 and 60 Months (intervention arms only)
  Type-2 diabetes status will be evaluated by measuring Hemoglobin A1c (HbA1c)
Change from Baseline Metabolic Syndrome Status | 42 and 60 Months (intervention arms only)
  Metabolic syndrome status will be evaluated by standard markers. Metabolic syndrome is defined as having at least three of the following:
  * Waist circumference: ≥40 inches (men) or ≥35 inches (women)
  * Fasting triglycerides: ≥150 mg/dL
  * HDL-C: <40 mg/dL (men) or <50 mg/dL (women)
  * Blood pressure: ≥130/85 mm Hg or use of hypertensive medication
  * Fasting glucose: ≥ 100 mg/dL or use of hyperglycemia medication
Change from Baseline Body Weight | 42 and 60 Months (intervention arms only)
  Body weight will be evaluated on a calibrated scale

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hallberg, DO, MS, Principal Investigator — Indiana University Health
Locations (1):
- IU Health Arnett Medical Weight Loss, West Lafayette, Indiana, United States

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity among adults: United States, 2011-2012. NCHS Data Brief. 2013 Oct;(131):1-8. PMID 24152742
- [Background] Flegal KM, Carroll MD, Ogden CL, Curtin LR. Prevalence and trends in obesity among US adults, 1999-2008. JAMA. 2010 Jan 20;303(3):235-41. doi: 10.1001/jama.2009.2014. Epub 2010 Jan 13. PMID 20071471
- [Background] Mozumdar A, Liguori G. Persistent increase of prevalence of metabolic syndrome among U.S. adults: NHANES III to NHANES 1999-2006. Diabetes Care. 2011 Jan;34(1):216-9. doi: 10.2337/dc10-0879. Epub 2010 Oct 1. PMID 20889854
- [Background] Petersen KF, Dufour S, Savage DB, Bilz S, Solomon G, Yonemitsu S, Cline GW, Befroy D, Zemany L, Kahn BB, Papademetris X, Rothman DL, Shulman GI. The role of skeletal muscle insulin resistance in the pathogenesis of the metabolic syndrome. Proc Natl Acad Sci U S A. 2007 Jul 31;104(31):12587-94. doi: 10.1073/pnas.0705408104. Epub 2007 Jul 18. PMID 17640906
- [Background] Volek JS, Phinney SD, Forsythe CE, Quann EE, Wood RJ, Puglisi MJ, Kraemer WJ, Bibus DM, Fernandez ML, Feinman RD. Carbohydrate restriction has a more favorable impact on the metabolic syndrome than a low fat diet. Lipids. 2009 Apr;44(4):297-309. doi: 10.1007/s11745-008-3274-2. Epub 2008 Dec 12. PMID 19082851
- [Background] Volek JS, Fernandez ML, Feinman RD, Phinney SD. Dietary carbohydrate restriction induces a unique metabolic state positively affecting atherogenic dyslipidemia, fatty acid partitioning, and metabolic syndrome. Prog Lipid Res. 2008 Sep;47(5):307-18. doi: 10.1016/j.plipres.2008.02.003. Epub 2008 Mar 15. PMID 18396172
- [Background] Volek JS, Feinman RD. Carbohydrate restriction improves the features of Metabolic Syndrome. Metabolic Syndrome may be defined by the response to carbohydrate restriction. Nutr Metab (Lond). 2005 Nov 16;2:31. doi: 10.1186/1743-7075-2-31. PMID 16288655
- [Background] Santos FL, Esteves SS, da Costa Pereira A, Yancy WS Jr, Nunes JP. Systematic review and meta-analysis of clinical trials of the effects of low carbohydrate diets on cardiovascular risk factors. Obes Rev. 2012 Nov;13(11):1048-66. doi: 10.1111/j.1467-789X.2012.01021.x. Epub 2012 Aug 21. PMID 22905670
- [Background] Bistrian BR, Blackburn GL, Flatt JP, Sizer J, Scrimshaw NS, Sherman M. Nitrogen metabolism and insulin requirements in obese diabetic adults on a protein-sparing modified fast. Diabetes. 1976 Jun;25(6):494-504. doi: 10.2337/diab.25.6.494. PMID 1278601
- [Background] Gumbiner B, Wendel JA, McDermott MP. Effects of diet composition and ketosis on glycemia during very-low-energy-diet therapy in obese patients with non-insulin-dependent diabetes mellitus. Am J Clin Nutr. 1996 Jan;63(1):110-5. doi: 10.1093/ajcn/63.1.110. PMID 8604657
- [Background] Dashti HM, Al-Zaid NS, Mathew TC, Al-Mousawi M, Talib H, Asfar SK, Behbahani AI. Long term effects of ketogenic diet in obese subjects with high cholesterol level. Mol Cell Biochem. 2006 Jun;286(1-2):1-9. doi: 10.1007/s11010-005-9001-x. Epub 2006 Apr 21. PMID 16652223
- [Background] Yancy WS Jr, Foy M, Chalecki AM, Vernon MC, Westman EC. A low-carbohydrate, ketogenic diet to treat type 2 diabetes. Nutr Metab (Lond). 2005 Dec 1;2:34. doi: 10.1186/1743-7075-2-34. PMID 16318637
- [Background] Nielsen JV, Joensson EA. Low-carbohydrate diet in type 2 diabetes: stable improvement of bodyweight and glycemic control during 44 months follow-up. Nutr Metab (Lond). 2008 May 22;5:14. doi: 10.1186/1743-7075-5-14. PMID 18495047
- [Background] Hussain TA, Mathew TC, Dashti AA, Asfar S, Al-Zaid N, Dashti HM. Effect of low-calorie versus low-carbohydrate ketogenic diet in type 2 diabetes. Nutrition. 2012 Oct;28(10):1016-21. doi: 10.1016/j.nut.2012.01.016. Epub 2012 Jun 5. PMID 22673594
- [Background] Action to Control Cardiovascular Risk in Diabetes Study Group; Gerstein HC, Miller ME, Byington RP, Goff DC Jr, Bigger JT, Buse JB, Cushman WC, Genuth S, Ismail-Beigi F, Grimm RH Jr, Probstfield JL, Simons-Morton DG, Friedewald WT. Effects of intensive glucose lowering in type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2545-59. doi: 10.1056/NEJMoa0802743. Epub 2008 Jun 6. PMID 18539917
- [Background] ADVANCE Collaborative Group; Patel A, MacMahon S, Chalmers J, Neal B, Billot L, Woodward M, Marre M, Cooper M, Glasziou P, Grobbee D, Hamet P, Harrap S, Heller S, Liu L, Mancia G, Mogensen CE, Pan C, Poulter N, Rodgers A, Williams B, Bompoint S, de Galan BE, Joshi R, Travert F. Intensive blood glucose control and vascular outcomes in patients with type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2560-72. doi: 10.1056/NEJMoa0802987. Epub 2008 Jun 6. PMID 18539916
- [Background] Seip RL, Volek JS, Windemuth A, Kocherla M, Fernandez ML, Kraemer WJ, Ruano G. Physiogenomic comparison of human fat loss in response to diets restrictive of carbohydrate or fat. Nutr Metab (Lond). 2008 Feb 6;5:4. doi: 10.1186/1743-7075-5-4. PMID 18254975
- [Background] Qi Q, Bray GA, Smith SR, Hu FB, Sacks FM, Qi L. Insulin receptor substrate 1 gene variation modifies insulin resistance response to weight-loss diets in a 2-year randomized trial: the Preventing Overweight Using Novel Dietary Strategies (POUNDS LOST) trial. Circulation. 2011 Aug 2;124(5):563-71. doi: 10.1161/CIRCULATIONAHA.111.025767. Epub 2011 Jul 11. PMID 21747052
- [Background] Zhang X, Qi Q, Zhang C, Smith SR, Hu FB, Sacks FM, Bray GA, Qi L. FTO genotype and 2-year change in body composition and fat distribution in response to weight-loss diets: the POUNDS LOST Trial. Diabetes. 2012 Nov;61(11):3005-11. doi: 10.2337/db11-1799. Epub 2012 Aug 13. PMID 22891219
- [Background] Gardner CD. Tailoring dietary approaches for weight loss. Int J Obes Suppl. 2012 Jul;2(Suppl 1):S11-S15. doi: 10.1038/ijosup.2012.4. PMID 25089189
- [Background] McClain AD, Otten JJ, Hekler EB, Gardner CD. Adherence to a low-fat vs. low-carbohydrate diet differs by insulin resistance status. Diabetes Obes Metab. 2013 Jan;15(1):87-90. doi: 10.1111/j.1463-1326.2012.01668.x. Epub 2012 Aug 22. PMID 22831182
- [Background] Bots ML, Hoes AW, Koudstaal PJ, Hofman A, Grobbee DE. Common carotid intima-media thickness and risk of stroke and myocardial infarction: the Rotterdam Study. Circulation. 1997 Sep 2;96(5):1432-7. doi: 10.1161/01.cir.96.5.1432. PMID 9315528
- [Background] Stein JH, Korcarz CE, Hurst RT, Lonn E, Kendall CB, Mohler ER, Najjar SS, Rembold CM, Post WS; American Society of Echocardiography Carotid Intima-Media Thickness Task Force. Use of carotid ultrasound to identify subclinical vascular disease and evaluate cardiovascular disease risk: a consensus statement from the American Society of Echocardiography Carotid Intima-Media Thickness Task Force. Endorsed by the Society for Vascular Medicine. J Am Soc Echocardiogr. 2008 Feb;21(2):93-111; quiz 189-90. doi: 10.1016/j.echo.2007.11.011. No abstract available. PMID 18261694
- [Background] Shimazu T, Hirschey MD, Newman J, He W, Shirakawa K, Le Moan N, Grueter CA, Lim H, Saunders LR, Stevens RD, Newgard CB, Farese RV Jr, de Cabo R, Ulrich S, Akassoglou K, Verdin E. Suppression of oxidative stress by beta-hydroxybutyrate, an endogenous histone deacetylase inhibitor. Science. 2013 Jan 11;339(6116):211-4. doi: 10.1126/science.1227166. Epub 2012 Dec 6. PMID 23223453
- [Background] Robroek SJ, van den Berg TI, Plat JF, Burdorf A. The role of obesity and lifestyle behaviours in a productive workforce. Occup Environ Med. 2011 Feb;68(2):134-9. doi: 10.1136/oem.2010.055962. Epub 2010 Sep 27. PMID 20876556
- [Derived] Lyman KS, Athinarayanan SJ, McKenzie AL, Pearson CL, Adams RN, Hallberg SJ, McCarter JP, Volek JS, Phinney SD, Andrawis JP. Continuous care intervention with carbohydrate restriction improves physical function of the knees among patients with type 2 diabetes: a non-randomized study. BMC Musculoskelet Disord. 2022 Mar 29;23(1):297. doi: 10.1186/s12891-022-05258-0. PMID 35351093
- [Derived] Athinarayanan SJ, Adams RN, Hallberg SJ, McKenzie AL, Bhanpuri NH, Campbell WW, Volek JS, Phinney SD, McCarter JP. Long-Term Effects of a Novel Continuous Remote Care Intervention Including Nutritional Ketosis for the Management of Type 2 Diabetes: A 2-Year Non-randomized Clinical Trial. Front Endocrinol (Lausanne). 2019 Jun 5;10:348. doi: 10.3389/fendo.2019.00348. eCollection 2019. PMID 31231311
- [Derived] Vilar-Gomez E, Athinarayanan SJ, Adams RN, Hallberg SJ, Bhanpuri NH, McKenzie AL, Campbell WW, McCarter JP, Phinney SD, Volek JS, Chalasani N. Post hoc analyses of surrogate markers of non-alcoholic fatty liver disease (NAFLD) and liver fibrosis in patients with type 2 diabetes in a digitally supported continuous care intervention: an open-label, non-randomised controlled study. BMJ Open. 2019 Feb 25;9(2):e023597. doi: 10.1136/bmjopen-2018-023597. PMID 30803948
- [Derived] Bhanpuri NH, Hallberg SJ, Williams PT, McKenzie AL, Ballard KD, Campbell WW, McCarter JP, Phinney SD, Volek JS. Cardiovascular disease risk factor responses to a type 2 diabetes care model including nutritional ketosis induced by sustained carbohydrate restriction at 1 year: an open label, non-randomized, controlled study. Cardiovasc Diabetol. 2018 May 1;17(1):56. doi: 10.1186/s12933-018-0698-8. PMID 29712560
- [Derived] Hallberg SJ, McKenzie AL, Williams PT, Bhanpuri NH, Peters AL, Campbell WW, Hazbun TL, Volk BM, McCarter JP, Phinney SD, Volek JS. Effectiveness and Safety of a Novel Care Model for the Management of Type 2 Diabetes at 1 Year: An Open-Label, Non-Randomized, Controlled Study. Diabetes Ther. 2018 Apr;9(2):583-612. doi: 10.1007/s13300-018-0373-9. Epub 2018 Feb 7. PMID 29417495